CLINICAL TRIAL: NCT01463540
Title: A Multicentric, Randomised Clinical Trial Comparing Short and Long Time Outcome of Gastrostomy Tube Placed After Gastropexy, Versus Gastrostomy Tube Placed Using the Traditional Push/Pull Techniques
Brief Title: Gastrostomy Tube Placed After Gastropexy Versus Gastrostomy Tube Placed Using the Traditional Push/Pull Techniques
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASMN1PEG
Record Dates: First submitted 2011-10-30; First posted 2011-11-02 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2015-08

CONDITIONS: Gastrostomy, Methods
Keywords: Enteral nutrition; Gastrostomy, adverse effects; Gastrostomy, nursing; Endoscopy,gastrointestinal; Surgical wound infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Push/pull endoscopic gastrostomy (Active Comparator)
  Interventions: Device: A 20 Fr gastrostomy tube, placed using push/pull techniques.
- Gastrostomy after gastropexy (Experimental)
  Interventions: Device: A 20 Fr balloon type tube, placed after gastropexy.

INTERVENTIONS:
Device: A 20 Fr gastrostomy tube, placed using push/pull techniques. — In this group a 20 Fr gastrostomy tube will be placed, of the type in use at each centre, using the push or the pull method. Positioning of the gastrostomy tube will be carried out endoscopically in sedated patients, after antibiotic prophylaxis. Single dose ampicillin/sulbactam 1g/500 mg will be infused intravenously 30 minutes before positioning. In patients just receiving antibiotic therapy, as treatment of concomitant disease, the current therapy will be continued and antibiotic prophylaxis with ampicillin/sulbactam will be not given.
  Arms: Push/pull endoscopic gastrostomy
Device: A 20 Fr balloon type tube, placed after gastropexy. — In this group a 20 Fr balloon type gastrostomy tube will be placed endoscopically, after gastropexy performed using the Kimberly Clarke MIC Introducer kit, according to the instructions suggested by the manufacturer. The kit includes 4 T-fasteners (only 3 are usually placed in clinical use) and a serial 24 Fr dilator with a pell-away sheath. All commercially available brands of balloon type gastrostomy tubes will be allowed for use in the study. Positioning of the gastrostomy tube will be carried out in sedated patients, after antibiotic prophylaxis (Single dose ampicillin/sulbactam 1g/500 mg ev.). In patients just receiving antibiotic therapy, as treatment of concomitant disease, the current therapy will be continued and antibiotic prophylaxis will be not given.
  Other Names: Kimberly Clark MIC Introducer Kit Product CODE 98423.
  Arms: Gastrostomy after gastropexy

SUMMARY:
Endoscopic placement of a percutaneous gastrostomy tube is a safe, efficient and well standardized technique. Two variants of this maneuver - the pull and the push techniques - are widespread worldwide. More recently different techniques, that allow the direct insertion of a gastrostomy tube has been described. The common characteristic shared by all these technique is the fact that the gastrostomy tube is inserted directly into the stomach (without passing through the pharynx), after the gastric and abdominal wall have been securely fasten together (gastropexy).

Advantage of direct techniques are the followings:

1. the tube can placed also in the case of an oesophageal stenosis
2. studies suggest that the peristomal wound infection are less frequent using direct techniques
3. in some variants of these techniques, a balloon type gastrostomy tube or a button can be placed also in the case of first positioning. Both the balloon type tube and the button are easy to be changed also at the bed-side.

Drawbacks of the direct techniques are:

1. these technique are easy, but a little more cumbersome than classic push or pull maneuvers
2. operators are often not familiar with direct insertion
3. kits suited for direct insertion are generally more costly than available kits for push or pull placement of gastrostomy tube.

The kit manufactured by the Kimberly-Clark (MIC Introducer kit) allows direct insertion of a balloon type gastrostomy tube or of a button and it is interesting, because it makes simple to perform the gastropexy.

The study aim is to confirm that the use of the Kit Introducer MIC, may allow safe placement of a gastrostomy tube and may reduce the incidence of peristomal wound infection. Furthermore if a balloon type gastrostomy tube or a button are positioned, they may be changed at the bed-side, without referral of the patient to the endoscopic unit or to an other sanitary facility.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients, candidates to percutaneous endoscopic gastrostomy placement for any common clinical indication, in the centres participating to the study.

Exclusion Criteria:

* age < 18
* age > 85 years old
* pregnancy
* coagulation deficit or anti-coagulant oral therapy
* total gastrectomy
* absence of trans-illumination, verified during esophagogastroduodenoscopy
* pharyngeal or esophageal stenosis, not allowing the passage of a standard scope;
* ascitis
* active gastric ulcer
* the patient or his tutor do not consent to the study
* documented allergy to penicillin
* ASA V.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of patients with peristomal wound infection. | From the date of randomization up to 30 days, or until the date of death from any cause, whichever came first.
  Peristomal wound infection is defined as Jain score > 8, or presence of purulent exudates.
Number of patients with major complication. | From the date of randomization up to 30 days, or until the date of death from any cause, whichever came first.
  Major complications include: 1. perforation/peritonitis or hemoperitoneum, requiring surgery; 2. Clinically relevant gastrointestinal bleeding (loss of more than 2g Hb during 24 hours and/or requiring transfusion and/or endoscopic or surgical treatment); 3. aspiration pneumonia; 4. Burried bumper syndrome.
Number of failures of positioning the gastrostomy tube. | From the start until the end of the endoscopic procedure.
  Gastrostomy tube positioning will be performed immediately after randomization.Patients will be randomised by the endoscopist, during EGD. Only one attempt of positioning the gastrostomy tube will be allowed. Further attempts of positioning a gastrostomy tube after a failure will be not relevant to the pourpose of the study. Failures do not include patients with uncorrect positioning of the tube, if the misplacement is diagnosed after the end of the endoscopic procedure.

SECONDARY OUTCOMES:
Mean Jain's score. | Jain score will be measured at follow up visits during the first month after positioning of the gastrostomy tube (on 7th, 15th, 30th days).
  Jain's score is a validated scoring system, proposed to evaluate peristomal infection.
Number of gastrostomy tube substitutions for each patient. | From date of randomization until the date of definitive removal of the tube or date of death from any cause, whichever came first, assessed up to 13 months.
  The setting of the substitution will be recorded (at bed site, endoscopic unit, other sanitary facilities).
Number of episodes of referral to the hospital or to any sanitary facility (outpatient clinic visit included), due to gastrostomy tube. | From date of randomization until the date of definitive removal of the tube or date of death from any cause, whichever came first, assessed up to 13 months
Days of antibiotic therapy after gastrostomy tube positioning. | From the date of randomization up to 30 days, or until the date of death from any cause, whichever came first.
Mean time required for tube positioning, as measured in minutes. | From the start until the end of the endoscopic procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Camellini, MD, Principal Investigator — Azienda USL Reggio Emilia - IRCCS; Vincenzo Mirante, MD, Study Chair — Nuovo Ospedale Estense - AUSL Modena; Veronica Iori, MD, Study Chair — Azienda USL Reggio Emilia - IRCCS; Angela Mazzocchi, MD, Study Chair — Artificial Nutrition Interdisciplinary Team - AUSL Reggio Emilia; Fabio Fabbian, MD, Study Chair — Endoscopy Unit - AUSL RE; Rita Conigliaro, MD, Study Chair — Nuovo Ospedale Estense - AUSL Modena; Romano Sassatelli, MD, Study Chair — Azienda USL Reggio Emilia - IRCCS; Giorgio Iori, Reg. Nurse, Study Chair — Azienda USL Reggio Emilia - IRCCS
Locations (3):
- Italy (3):
  - Digestive Endoscopy Unit - Nuovo Ospedale Estense, Modena, MO
  - Gastroenterology and Digestive Endoscopy Unit - Arcispedale Santa Maria Nuova, Reggio Emilia, RE
  - Endoscopic Unit "South Area" - AUSL Reggio Emilia, Scandiano, RE

REFERENCES:
- [Background] Maetani I, Tada T, Ukita T, Inoue H, Sakai Y, Yoshikawa M. PEG with introducer or pull method: a prospective randomized comparison. Gastrointest Endosc. 2003 Jun;57(7):837-41. doi: 10.1016/s0016-5107(03)70017-0. PMID 12776029
- [Background] Jain NK, Larson DE, Schroeder KW, Burton DD, Cannon KP, Thompson RL, DiMagno EP. Antibiotic prophylaxis for percutaneous endoscopic gastrostomy. A prospective, randomized, double-blind clinical trial. Ann Intern Med. 1987 Dec;107(6):824-8. doi: 10.7326/0003-4819-107-6-824. PMID 3318609
- [Background] Shastri YM, Hoepffner N, Tessmer A, Ackermann H, Schroeder O, Stein J. New introducer PEG gastropexy does not require prophylactic antibiotics: multicenter prospective randomized double-blind placebo-controlled study. Gastrointest Endosc. 2008 Apr;67(4):620-8. doi: 10.1016/j.gie.2007.10.044. PMID 18374024
- [Background] Horiuchi A, Nakayama Y, Tanaka N, Fujii H, Kajiyama M. Prospective randomized trial comparing the direct method using a 24 Fr bumper-button-type device with the pull method for percutaneous endoscopic gastrostomy. Endoscopy. 2008 Sep;40(9):722-6. doi: 10.1055/s-2008-1077490. Epub 2008 Sep 4. PMID 18773341